CLINICAL TRIAL: NCT07252700
Title: Preventing Diabetes: Impact of an EMR-Based Intervention for Enhanced Pre-Diabetes Management in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lynette Goh (Other)
Collaborators: National University Health System, Singapore (Other); National University of Singapore (Other)
Responsible Party: Sponsor-Investigator, Lynette Goh, Senior Principal Dietitian, National University Polyclinics, Singapore
Organization: National University Polyclinics, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECOS Ref No.: 2025-1224
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pre Diabetes; Diabetes (DM)
Keywords: prediabetes; primary care; electronic medical records (EMR); OurPractice Advisories
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR-Based Intervention - Practice advisories (OPA) in electronic medical records (EMR) (Active Comparator): To implement a non-intrusive OPA in EMR (Epic) to appear in the OPA section of the Visit Navigator in Epic that will be triggered for patients with prediabetes to remind clinicians to fulfil the clinical workflow for managing patients with prediabetes
  Interventions: Behavioral: Electronic Medical Record-Based Clinical Decision Support
- Comparison Group (No Intervention): Control clinics continue to use the clinical workflow without EMR-based OPAs, representing usual care.

INTERVENTIONS:
Behavioral: Electronic Medical Record-Based Clinical Decision Support — A non-intrusive OurPractice Advisories (OPA) will be implemented in the Epic EMR system. The OPA will appear in the Visit Navigator and will be automatically triggered for patients with pre-diabetes. It will provide clinicians with reminders and decision-support options to complete the recommended clinical workflow for pre-diabetes management, including referrals, follow-up scheduling, HbA1c testing, and medication initiation when indicated.
  Arms: EMR-Based Intervention - Practice advisories (OPA) in electronic medical records (EMR)

SUMMARY:
The goal of this study is to find out if adding electronic medical record (EMR) prompts helps prevent people with pre-diabetes from developing diabetes. It will also look at how these prompts affect doctor and patient behaviors.

The main questions are:

Does it improve follow-up care, such as blood tests, referrals, and medication? Does the EMR prompt reduce the number of patients who progress to diabetes within six months?

Researchers will compare clinics that use EMR prompts with clinics that do not.

Participants will:

Receive usual care for pre-diabetes at their polyclinic In some clinics, doctors will see EMR prompts suggesting tests, referrals, and medication Complete surveys about their health and lifestyle at different time points

DETAILED DESCRIPTION:
This is a two-year cluster-randomized controlled trial conducted across eight primary care polyclinics within the National University Polyclinics (NUP) network in Singapore. These clinics provide multidisciplinary family medicine and chronic disease management services to a large and diverse population. All sites use a unified Electronic Medical Record (EMR) system (Epic, National University Health System cluster), which supports standardized clinical workflows, integrates decision-support tools, and enables secure extraction of de-identified data for research.

The study targets adults aged 21-59 years with prediabetes. All clinicians in both intervention and control clinics will receive standardized clinical training on updated prediabetes clinical practice guidelines and patient education materials. The updated workflow emphasizes lifestyle modification and behavioural counselling as the foundation of diabetes prevention. Clinicians are guided to refer patients to a dietitian or structured lifestyle programme if body mass index (BMI) is 23 kg/m² or above, counsel patients on nutrition and physical activity, schedule a six-month follow-up review, order HbA1c testing prior to the next review, and consider metformin initiation if HbA1c exceeds 6.5% after six months of lifestyle intervention, particularly in adults under 60 years with BMI ≥ 23 kg/m². Training will be conducted virtually during protected lunchtime sessions.

The study consists of three sequential phases. Phase 0 (Baseline) involves no workflow intervention, during which baseline EMR and survey data are collected. Phase 1 (Workflow Phase) introduces the standardized prediabetes clinical workflow across all clinics. Phase 2 (Prompt Phase) introduces EMR-based smart-set prompts only in intervention clinics to evaluate whether prompts further increase referrals, follow-up scheduling, HbA1c testing, and metformin prescribing beyond the workflow alone. Control clinics continue to use the standardized workflow without EMR prompts. The smart-set prompts are designed to be non-intrusive and provide decision support without interrupting workflow or overriding clinical judgment. Clinicians retain full autonomy to accept, modify, or dismiss suggested actions.

A sub-sample of approximately 300 patients will complete questionnaires assessing lifestyle behaviours and patient activation using the Consumer Health Activation Index (CHAI) to complement EMR-derived outcomes. Approximately 80-100 clinicians are expected to complete voluntary, anonymous surveys assessing knowledge, confidence, and clinical behaviours using the COM-B framework. Baseline clinical and survey data will be collected prior to intervention implementation, with follow-up data collected at multiple time points to evaluate short- and longer-term outcomes.

Intervention components include standardized workflow implementation and clinician education across all clinics, with additional EMR-based prompts implemented only in intervention clinics. Smart-set prompts integrated within Epic display automated reminders at the point of care, with options to facilitate orders for laboratory tests, referrals, medications, and follow-up scheduling. Prompts are non-mandatory to preserve clinician autonomy. The intervention is informed by the COM-B model to enhance clinician capability (through training and guidelines), opportunity (through EMR-enabled workflows and referral pathways), and motivation (through feedback and reinforcement). The Transtheoretical Model (TTM) will be used to monitor stages of change among both patients and clinicians.

Survey data will be collected electronically using FormSG, a secure, government-hosted platform approved for research use. All study data will be stored on institution-approved, PDPA-compliant servers with access restricted to authorized study personnel. Identifiable and de-identified datasets will be stored separately. De-identified datasets will be transferred to analysts using encrypted, password-protected channels. Only the Principal Investigator will have access to the linkage file containing study identifiers and personal identifiers. Hard-copy consent forms will be stored in locked cabinets accessible only to the Principal Investigator. Study data will be retained for six years following study completion in accordance with institutional policy, after which electronic data will be securely deleted and physical records destroyed.

Analyses will follow the intention-to-treat principle, with participants analysed according to their assigned clinic groups. Baseline characteristics will be summarized descriptively. Changes over time and differences between intervention and control clinics will be examined using regression models appropriate to outcome type, including mixed-effects logistic regression to account for clustering at the clinic level. Time-to-event analyses using Cox proportional hazards regression will be used to assess progression to diabetes while accounting for variable follow-up durations. Missing data will be addressed using multiple imputation, and sensitivity analyses will be conducted to assess robustness of findings. All analyses will use two-sided tests with a significance level of 0.05.

Outcome data will be collected at baseline, 6 months, 12 months, and at 18 and 24 months to assess short- and longer-term effects of workflow and EMR-based decision-support implementation.

This study will contribute evidence on the effectiveness of a non-intrusive, EMR-embedded clinical decision-support system for improving guideline-concordant prediabetes care in primary care and inform scalable strategies for diabetes prevention.

ELIGIBILITY:
Inclusion Criteria for study population (EMR based analytic cohort):

* All adults aged 21 to 59 years with prediabetes who attend any of the eight participating polyclinics during the study period will be included in the EMR-based analytic cohort.
* Prediabetes is defined as impaired fasting glucose or impaired glucose tolerance according to standard clinical criteria, with either diagnosis documented in the EMR problem list or visit diagnosis.
* Individuals with a prior diagnosis of diabetes will be excluded.

Inclusion Criteria for patient surveys:

* Adults aged 40-59 years
* Diagnosed with prediabetes (impaired fasting glucose or impaired glucose tolerance)
* Receiving routine follow-up care at NUP polyclinics
* Able to provide written informed consent
* Able to complete questionnaires in English

Exclusion criteria for patient surveys:

* Prior diagnosis of diabetes mellitus or gestational diabetes
* Severe acute or chronic liver or kidney disease
* Pregnancy
* Cognitive impairment
* Inability to communicate in English

Inclusion Criteria for clinician surveys:

* All clinicians that consult patients in National University Polyclinics
* No exclusion criteria specified for clinicians

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Guideline-concordant prediabetes care | From enrollment to the end of intervention period at 24 months. collected at baseline, 6 months, 12, months, 18 months and 24 months.
  The primary outcome of this study is the proportion of patients receiving guideline-concordant prediabetes care within 6 months of the index consultation, defined as the first prediabetes consultation during the study period at which patient meets eligibility criteria for prediabetes.
  1. HbA1c test ordered and recorded in the EMR.
  2. Referral to a dietitian or structured lifestyle programme placed and recorded in the EMR.
  3. Follow-up visit ordered by the attending clinician.
  4. Metformin prescription recorded in the EMR for eligible patients (HbA1c ≥ 6.5%).
  Scale: Guideline-concordant care is defined as a composite measure in which patients have at least two of the following four clinician-initiated care processes captured in EMR data:
  Method: EMR data extracted from the Epic system, including laboratory orders, referrals, visit scheduling, and medication prescriptions.

SECONDARY OUTCOMES:
Progression to Diabetes | Up to 24 months after index consultation
  Progression from prediabetes to diabetes at 6, 12, 18 and 24 months. Diabetes will be defined according to the Agency for Care Effectiveness (ACE) Appropriate Care Guide as fasting plasma glucose ≥7.0 mmol/L, HbA1c ≥7.0%, or 2-hour plasma glucose ≥11.1 mmol/L during an oral glucose tolerance test, as recorded in the EMR.
  Scale: Progression to diabetes, defined as the occurrence of diabetes during follow-up among patients with prediabetes at baseline.
  Method: Data extraction from EMR records
Patient health activation | Baseline, 6 months, and 12 months.
  Measured using the Consumer Health Activation Index (CHAI) questionnaire. Scores reflect patients' knowledge, skills, and confidence in managing their health. Minimum value: 10 Maximum value: 60. This will then be transformed into a 0 to 100 scale.
  Interpretation: Higher scores indicate greater activation. Method: Surveys administered to a sub-sample of approximately 300 patients
Clinician perceptions and satisfaction with the EMR-based intervention | Baseline, 6 months and 12 months
  Clinician perceptions and satisfaction with the EMR-based intervention will be assessed through an anonymous survey.
  Description: Survey assessing clinician confidence, familiarity with guidelines, current practices, use of EMR tools, and satisfaction with intervention. Includes multiple-choice and Likert-scale questions (4-point confidence/familiarity scales, 5-point frequency scales, 4-point agreement scales).
  Key areas:
  Clinician capability (knowledge, skills, confidence) Current practices in pre-diabetes management Use and integration of EMR tools Perceived barriers Impact of EMR tools on care delivery Overall satisfaction
  Interpretation: Responses will be analyzed individually and in aggregate to assess changes in clinician perceptions, practices, and satisfaction over time. Higher scores on agreement scales generally indicate more positive perceptions or greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Privacy and Confidentiality: Our study involves some sensitive health information. Even with de-identification, there remains a risk of re-identification, particularly given the detailed nature of our data and the specific population studied.
  Ethical Constraints: Our informed consent process and ethics approval did not explicitly include provisions for broad data sharing beyond the immediate research team and oversight committees.
  Regulatory Compliance: Local health data protection regulations place strict limitations on the sharing of individual-level health data, even in anonymized form.
  However, we are committed to scientific transparency and reproducibility. Therefore, we will make aggregate data, statistical codes, and detailed study protocols available upon reasonable request, subject to approval by our institutional review board and data access committee.

REFERENCES:
- [Background] Wolf MS, Smith SG, Pandit AU, Condon DM, Curtis LM, Griffith J, O'Conor R, Rush S, Bailey SC, Kaplan G, Haufle V, Martin D. Development and Validation of the Consumer Health Activation Index. Med Decis Making. 2018 Apr;38(3):334-343. doi: 10.1177/0272989X17753392. Epub 2018 Feb 13. PMID 29436308
- [Background] Goh SY, Ang SB, Bee YM, Chen YT, Gardner DS, Ho ET, Adaikan K, Lee YC, Lee CH, Lim FS, Lim HB, Lim SC, Seow J, Soh AW, Sum CF, Tai ES, Thai AC, Wong TY, Yap F. Ministry of Health Clinical Practice Guidelines: Diabetes Mellitus. Singapore Med J. 2014 Jun;55(6):334-47. doi: 10.11622/smedj.2014079. PMID 25017409
- [Background] Shuyu Ng C, Toh MP, Ko Y, Yu-Chia Lee J. Direct medical cost of type 2 diabetes in singapore. PLoS One. 2015 Mar 27;10(3):e0122795. doi: 10.1371/journal.pone.0122795. eCollection 2015. PMID 25816299
- [Background] Ang YG, WU CX, Toh MP, Chia KS, Heng BH. Progression rate of newly diagnosed impaired fasting glycemia to type 2 diabetes mellitus: a study using the National Healthcare Group Diabetes Registry in Singapore. J Diabetes. 2012 Jun;4(2):159-63. doi: 10.1111/j.1753-0407.2011.00169.x. PMID 22059651
- [Background] Tomic D, Shaw JE, Magliano DJ. The burden and risks of emerging complications of diabetes mellitus. Nat Rev Endocrinol. 2022 Sep;18(9):525-539. doi: 10.1038/s41574-022-00690-7. Epub 2022 Jun 6. PMID 35668219
- [Background] Saito T, Watanabe M, Nishida J, Izumi T, Omura M, Takagi T, Fukunaga R, Bandai Y, Tajima N, Nakamura Y, Ito M; Zensharen Study for Prevention of Lifestyle Diseases Group. Lifestyle modification and prevention of type 2 diabetes in overweight Japanese with impaired fasting glucose levels: a randomized controlled trial. Arch Intern Med. 2011 Aug 8;171(15):1352-60. doi: 10.1001/archinternmed.2011.275. PMID 21824948
- [Background] Keck JW, Roper KL, Hieronymus LB, Thomas AR, Huang Z, Westgate PM, Fowlkes JL, Cardarelli R. Primary Care Cluster RCT to Increase Diabetes Prevention Program Referrals. Am J Prev Med. 2020 Jul;59(1):79-87. doi: 10.1016/j.amepre.2020.02.008. Epub 2020 May 14. PMID 32418801
- [Background] Jiang Q, Li JT, Sun P, Wang LL, Sun LZ, Pang SG. Effects of lifestyle interventions on glucose regulation and diabetes risk in adults with impaired glucose tolerance or prediabetes: a meta-analysis. Arch Endocrinol Metab. 2022 Apr 28;66(2):157-167. doi: 10.20945/2359-3997000000441. Epub 2022 Mar 14. PMID 35289514
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Lim RBT, Wee WK, For WC, Ananthanarayanan JA, Soh YH, Goh LML, Tham DKT, Wong ML. Health education and communication needs among primary care patients with prediabetes in Singapore: A mixed methods approach. Prim Care Diabetes. 2020 Jun;14(3):254-264. doi: 10.1016/j.pcd.2019.08.008. Epub 2019 Sep 23. PMID 31558372
- [Background] Cheah MH, Goh LH, Zheng RM, Burkill S, Young DYL. Prediabetes guidelines adherence and health outcomes at a Singapore primary health care institution. Singapore Med J. 2024 Jan 8. doi: 10.4103/singaporemedj.SMJ-2021-220. Online ahead of print. No abstract available. PMID 38189477
- [Background] Holliday CS, Williams J, Salcedo V, Kandula NR. Clinical Identification and Referral of Adults With Prediabetes to a Diabetes Prevention Program. Prev Chronic Dis. 2019 Jun 27;16:E82. doi: 10.5888/pcd16.180540. PMID 31255186
- [Background] Lessing SE, Hayman LL. Diabetes Care and Management Using Electronic Medical Records: A Systematic Review. J Diabetes Sci Technol. 2019 Jul;13(4):774-782. doi: 10.1177/1932296818815507. Epub 2018 Dec 17. PMID 30556418
- [Background] O'Connor PJ, Crain AL, Rush WA, Sperl-Hillen JM, Gutenkauf JJ, Duncan JE. Impact of an electronic medical record on diabetes quality of care. Ann Fam Med. 2005 Jul-Aug;3(4):300-6. doi: 10.1370/afm.327. PMID 16046561
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Meigs JB, Cagliero E, Dubey A, Murphy-Sheehy P, Gildesgame C, Chueh H, Barry MJ, Singer DE, Nathan DM. A controlled trial of web-based diabetes disease management: the MGH diabetes primary care improvement project. Diabetes Care. 2003 Mar;26(3):750-7. doi: 10.2337/diacare.26.3.750. PMID 12610033
- [Background] Gerstein HC, Santaguida P, Raina P, Morrison KM, Balion C, Hunt D, Yazdi H, Booker L. Annual incidence and relative risk of diabetes in people with various categories of dysglycemia: a systematic overview and meta-analysis of prospective studies. Diabetes Res Clin Pract. 2007 Dec;78(3):305-12. doi: 10.1016/j.diabres.2007.05.004. Epub 2007 Jun 29. PMID 17601626
- [Background] Phan TP, Alkema L, Tai ES, Tan KH, Yang Q, Lim WY, Teo YY, Cheng CY, Wang X, Wong TY, Chia KS, Cook AR. Forecasting the burden of type 2 diabetes in Singapore using a demographic epidemiological model of Singapore. BMJ Open Diabetes Res Care. 2014 Jun 11;2(1):e000012. doi: 10.1136/bmjdrc-2013-000012. eCollection 2014. PMID 25452860
- See also: National population health survey 2024 — https://www.hpb.gov.sg/docs/default-source/pdf/nphs-2024-survey-report.pdf